CLINICAL TRIAL: NCT03406013
Title: True NTH Community of Wellness Internet-Based Exercise and Diet Support for Prostate Cancer Survivors
Brief Title: Internet-Based Exercise and Diet Support in Prostate Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Movember Foundation (Other)
Responsible Party: Principal Investigator, Kerri Winters, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00016703; NCI-2017-01048 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00016703 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2017-07-22; First posted 2018-01-23 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Cancer Survivor; Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prescriptions; Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (Active Comparator): Written Information
  Interventions: Behavioral: Written Information
- Group II (Experimental): Written Information Prescription
  Interventions: Behavioral: Written Information; Behavioral: Prescription
- Group III (Experimental): Written Information Prescription Technology
  Interventions: Behavioral: Written Information; Behavioral: Prescription; Behavioral: Technology
- Group IV (Experimental): Written Information Prescription Technology Coaching
  Interventions: Behavioral: Written Information; Behavioral: Prescription; Behavioral: Technology; Behavioral: Coaching

INTERVENTIONS:
Behavioral: Written Information — Receive written information on diet and exercise relevant to older men with prostate cancer
Behavioral: Prescription — Participants receive tailored exercise prescription and tailored diet recommendations
  Arms: Group II; Group III; Group IV
Behavioral: Technology — Participants receive motivational text messages and can electronically log and track their exercise and diet habits
  Arms: Group III; Group IV
Behavioral: Coaching — Participants receive access to an exercise and diet coach to provide advice by phone and/or email
  Arms: Group IV

SUMMARY:
This pilot clinical trial studies how well the True NTH Community of Wellness internet-based exercise and diet support works in improving diet and exercise habits in prostate cancer survivors. Internet-based exercise and diet support may help better control treatment-related side effects and symptoms, better overall quality of life, and lower risk factors associated with cancer progression.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and acceptability of the Community of Wellness web portal among prostate cancer survivors by conducting a randomized controlled study comparing four levels of web-based content and interaction with participants.

SECONDARY OBJECTIVES:

I. To compare efficacy of four levels of web-based content in the Community of Wellness web portal in a pilot randomized controlled trial on exercise and dietary habits, self-efficacy for behavior change, motivation for exercise, and changes in treatment-related side effects.

OUTLINE: Patients are assigned to 1 of 4 groups.

GROUP I: Patients receive "Written Information" which includes access to the TrueNTH open access portal that provides basic written information about exercise and diet.

GROUP II: Patients receive access to "Written Information + Prescription", including written information plus additional an exercise prescription and tailored diet recommendations.

GROUP III: Patients receive access to "Written Information + Prescription + Technology", including written information, exercise prescription + diet recommendation and additional technology components. Patients complete diet and exercise behavior logs and receive educational and motivational text messages about healthy diet and exercise habits.

GROUP IV: Patients receive access to "Written Information + Prescription + Technology + Coaching" and receive written information, exercise prescription + diet recommendation, technology support and a 30-minute (each) diet and exercise consultation plus the ability to receive ongoing advice from coaches via the web portal.

After completion of intervention, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported prostate cancer diagnosis
* Able to read English on a computer screen
* Able to access a computer, tablet or smartphone at home or public location
* Access to a device capable of receiving plain text messages
* A personal email address

Exclusion Criteria:

* Men who have contraindications to exercise based the American College of Sports Medicine 2016 Exercise pre-participation screening criteria and who do not receive a physician clearance to participate in the moderate intensity physical activity with one or more of the following self-reported conditions:

  * heart attack
  * heart surgery, cardiac catheterization, or coronary angioplasty
  * pacemaker/implantable cardiac defibrillator/rhythm disturbance
  * heart valve disease
  * heart failure
  * heart transplantation
  * congenital heart disease
  * diabetes
  * kidney (renal) disease
  * chest discomfort with exertion
  * unreasonable breathlessness
  * dizziness, fainting or blackouts
  * ankle swelling
  * unpleasant awareness of forceful, rapid or irregular heart rate
  * burning or cramping sensations in your lower legs when walking short distance

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Accrual success | Up to 3 months
  Measured as ability to recruit target sample size within one year
Retention | Up to 6 months
  Measured as the % of men who complete post-intervention and follow-up measures out of the total # of men enrolled
Adherence to the study | Up to 3 months
  Measured as the # of times that a man visits the portal over three months

SECONDARY OUTCOMES:
Community Healthy Activities Model Program for Seniors (CHAMPS) physical activity survey | Baseline, 3 months, and 6 months
  CHAMPS estimates total weekly energy expenditure (in kilocalories per week) from low to vigorous intensity physical activities for older adults.
Harvard T.H. Chan School of Public Health Food Frequency Questionnaire for adults from 2007 | Baseline, 3 months, and 6 months
  This 132-item survey assesses dietary intake over the past month in categories from "never or less than once per month" to "6 or more times per day" and supports examining major food and nutrient categories of the U.S. diet.
Self-Efficacy for Exercise | Baseline, 3 months, and 6 months
  A 6-item measure of Self-efficacy for Exercise will be used. Summed scores range from 6-30, and higher scores indicate higher self-efficacy.
Physical Activity Stage Assessment | Baseline, 3 months, and 6 months
  This 5-question measure asks the person to select one description, from a choice of five, which describes his current activity behavior.
Charlson Comorbidity Index | Baseline, 3 months, and 6 months
  The Charlson Comorbidity Index is a weighted index to predict mortality. Scores range from 0-37, with higher scores indicating more chronic medical conditions.
Self-Efficacy for Diet | Baseline, 3 months, and 6 months
  Diet self-efficacy will be measured by having participants rate their confidence in performing each recommended task (e.g., two more servings of cooked tomatoes per week) using a Likert scale.
Pittsburgh Sleep Quality Index | Baseline, 3 months, and 6 months
  This self-report questionnaire assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score.
Memorial Anxiety Scale for Prostate Cancer (MAX-PC) | Baseline, 3 months, and 6 months
  MAX-PC is an 18 item scale to facilitate the identification and assessment of men with prostate cancer-related anxiety. This scale consists of three subscales that measure general prostate cancer anxiety, anxiety related to prostate specific antigen (PSA) levels in particular, and fear of recurrence.
PROMIS 7-item Short Form - Fatigue | Baseline, 3 months, and 6 months
  PROMIS - Fatigue evaluates self-reported symptoms of fatigue, from mild subjective feelings of tiredness to an overwhelming sense of exhaustion over the past seven days.
Behavioral Regulation in Exercise Questionnaire (BREQ2) | Baseline, 3 months, and 6 months
  BREQ2 measures the continuum of behavioral regulation in exercise psychology research. This questionnaire concerns the reasons why a person exercises regularly, works out, or engages in other such physical activities. It is structured so that it asks one question and provides responses that represent external regulation, introjected regulation, identified regulation, and intrinsic motivation.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Baseline, 3 months, and 6 months
  EORTC QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients and has five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status / QoL scale, and a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnea, loss of appetite, insomnia, constipation and diarrhea) and perceived financial impact of the disease. Scores range from 0-100, with higher functional scale scores indicating a higher level of healthy functioning while a higher score for a symptom scale represents a higher level of symptomatology or problems.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Winters-Stone, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Oregon Health & Science University, Portland, Oregon

REFERENCES:
- [Derived] Chan JM, Van Blarigan EL, Langlais CS, Zhao S, Ramsdill JW, Daniel K, Macaire G, Wang E, Paich K, Kessler ER, Beer TM, Lyons KS, Broering JM, Carroll PR, Kenfield SA, Winters-Stone KM. Feasibility and Acceptability of a Remotely Delivered, Web-Based Behavioral Intervention for Men With Prostate Cancer: Four-Arm Randomized Controlled Pilot Trial. J Med Internet Res. 2020 Dec 31;22(12):e19238. doi: 10.2196/19238. PMID 33382378
- [Derived] Winters-Stone KM, Kenfield SA, Van Blarigan EL, Moe EL, Ramsdill JW, Daniel K, Macaire G, Paich K, Kessler ER, Kucuk O, Gillespie TW, Lyons KS, Beer TM, Broering JM, Carroll PR, Chan JM. Effect of Increasing Levels of Web-Based Behavioral Support on Changes in Physical Activity, Diet, and Symptoms in Men With Prostate Cancer: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Nov 15;7(11):e11257. doi: 10.2196/11257. PMID 30442638